CLINICAL TRIAL: NCT04352504
Title: Clinical Trial to Determine the Efficacy of Almonds for Skin Radiance, Inflammation and Aging in Asian Females: A Pilot Study
Brief Title: The Effect of a Healthy Snack on Radiance, Aging and Inflammation of the Skin
Acronym: AlmondSkin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Almond Board of California (Other)
Responsible Party: Principal Investigator, Zhaoping Li, Professor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18-002001
Record Dates: First submitted 2020-04-09; First posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Skin Laxity
Keywords: skin; aging; almonds
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Intervention Model Description: This study will be a randomized, parallel group comparison of almonds vs. isocaloric pretzels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Almonds (Experimental): Consume 1.5 oz. serving almonds (246 calories) daily for 12 weeks
  Interventions: Other: Almond
- Pretzels (Active Comparator): Consume 2 oz. serving pretzels (216 calories) daily for 12 weeks
  Interventions: Other: Pretzel

INTERVENTIONS:
Other: Almond — Consume 1.5 oz. serving almonds (246 calories) daily for 12 weeks
  Arms: Almonds
Other: Pretzel — Consume 2 oz. serving of pretzels (216 calories) daily for 12 weeks
  Arms: Pretzels

SUMMARY:
The anti-oxidative and anti-inflammatory effects of polyphenolic compounds of almonds have been reported in limited animal studies and may have the potential to improve skin radiance. However, the skin related beneficial properties of almonds have not been investigated in humans. This study will examine the effects of almond consumption on human skin radiance in Asian women as a pilot.

DETAILED DESCRIPTION:
This study is a randomized, parallel group comparison of almonds vs. isocaloric pretzels carried out in accordance with the guidelines of the Human Subjects Protection Committee of the University of California, Los Angeles. All subjects will give written informed consent before the study begins. Subjects will consume 1.5 serving of almonds (~ 1.5 oz/d for 246kcal) or isocaloric pretzels (~ 2.0 oz/d for 216kcal) daily for 12 weeks and will undergo skin assessment at weeks 0, 4, 8 and 12. The assessments include skin radiance, sebum, and hydration/moisture. In addition the study will evaluate the effect of almond consumption on skin inflammation and aging by assessing UV-induced changes. Each group will have 20 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Asian females age 18-50 years' old (inclusive)
* Typically consume low fiber/polyphenol diet (beige diet)
* In good health with a BMI of 22 to 30 kg/ m2 (inclusive)
* Non-smokers
* Fitzpatrick Skin type II-IV
* Willing to maintain their normal skin care pattern for the duration of the study
* Willing to maintain their normal diet for the duration of the study but avoid almonds and pretzels.
* Subjects must read and sign the Institutional Review Board-approved written informed consent prior to the initiation of any study specific procedures or enrollment. A subject will be excluded for any condition that might compromise the ability to give truly informed consent.

Exclusion Criteria:

* Eating a high fiber/polyphenol diet or taking any medication or dietary supplement which interfere with the absorption of polyphenols.
* Women who are pregnant, lactating or trying to become pregnant.
* Currently taking any skin related prescription medication or supplements for less than 3 months.
* Currently consuming >14 alcoholic drinks (1 drink = 12 fl oz beer, 4 fl oz wine or 1.5 fl oz liquor) per week and/or unwilling to limit intake to less than 3 drinks per week during study participation or history of alcohol dependency.
* Screening laboratory value outside of the laboratory normal range that is considered clinically significant for study participation by the investigator.
* History or current diagnosis of serious medical condition such as Type I or Type II diabetes, major surgery, thyroid disease, heart problems (e.g. angina, bypass surgery, myocardial infarction, etc.), presence of implanted cardiac defibrillator or pacemaker, uncontrolled hypertension/high blood pressure, gastrointestinal disorders including chronic malabsorptive conditions, peptic ulcer disease, Crohn's disease, chronic diarrhea or active gallbladder disease, inflammatory bowel disease, fatty liver or cancer.
* Known allergy to almonds.
* Participation in another clinical trial within 30 days prior to enrollment.
* Any known clinically significant food allergy or intolerance.
* Currently taking any prescription medication or supplements for less than 3 months.
* Is unable or unwilling to comply with the study protocol.
* Subjects who cannot avoid excessive exposure to either natural or artificial sunlight.
* Received a nasally-delivered steroid, antibiotics within the past 14 days.
* Used topical antibiotic or topical steroid on the face,currently taking any prescription medications that increase the risk of photosensitivity or history of taking such medications in the less than 3 months (e.g. alpha-hydroxy acids in cosmetics, antibiotics (ciprofloxacin, doxycycline, levofloxacin, ofloxacin, tetracycline, trimethoprim), antifungals (flucytosine, griseofulvin, voriconazole), antihistamines (cetirizine, diphenhydramine, loratadine, promethazine, cyproheptadine)
* Subjects with a significant medical history or concurrent condition that the investigator(s) feel is not safe for the study
* Is unable or unwilling to comply with the study protocol.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
Skin radiance | 12 weeks
  Determine the clinical efficacy of almond consumption on skin radiance. The main criteria will be evaluated by clinical scoring using the coloring, luminosity, brightness, and transparency (C.L.B.T.TM)(18) scale and imperfections scale (dark circles, redness/rosacea, spots, and heterogeneity). The C.L.B.T.TM methodology allows assessing different descriptors of the complexion: coloring, luminosity, brightness, and transparency of facial skin.

SECONDARY OUTCOMES:
UV radiation sensitivity | 12 weeks
  Evaluate the effect of almond consumption on skin inflammation and aging by assessing UV-induced changes. This will done using the smallest dose of UV-B radiation capable of inducing erythema (minimal erythema dose [MED]). The minimal erythema dose (MED) is determined for each subject before (week 0) and after (week 12) the intervention. Prior to testing, the skin type will be evaluated based on the Fitzpatrick Skin Type scale. Participants with Fitzpatrick skin type 2-4 were included in the study and assessed for differences in their response to UV-B induced skin changes before and after 12 weeks of study intervention.
Skin aging (elasticity, sebum, and hydration/moisture) | 12 weeks
  Assess the effect of almond consumption on skin biological characteristics of elasticity, sebum, and hydration/moisture content using the Cutometer® Skin Elasticity Meter 580 (Courage and Khazaka Electronic GmbH, Cologne, Germany). The Cutometer measures the vertical deformation of the skin in millimeters when the skin is pulled by means of a controlled vacuum into the circular aperture, 6 mm in diameter, of the probe. In its standard configuration, the Cutometer is equipped with a measuring probe with a 2 mm aperture because the device is originally designed to measure only the elastic properties of the epidermis. Skin hydration will measured using the moisture/hydration probe that attaches to the Cutometer. The six sites measured include: forehead, under the eye, frontal cheek, crow's foot, lateral cheek, and inner forearm.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Center for Human Nutrition, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No